CLINICAL TRIAL: NCT00564551
Title: Impact of High Milk Product and Calcium Intake During Weight Loss on Markers of Insulin Resistance
Brief Title: Effect of Increased Intake of Low Fat Dairy Products on Weight Loss and Insulin Resistance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Raylene Reimer, Associate Professor, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UC 21076
Record Dates: First submitted 2007-11-26; First posted 2007-11-28 (Estimated); Last update posted 2010-01-21 (Estimated); Status verified 2010-01

CONDITIONS: Impaired Glucose Tolerance; Type 2 Diabetes; Metabolic Syndrome
Keywords: Prediabetes; Type 2 diabetes; Metabolic syndrome; Insulin resistance syndrome; Weight loss; Milk products; Calcium
MeSH Terms: conditions — Glucose Intolerance; Diabetes Mellitus, Type 2; Metabolic Syndrome; Prediabetic State; Weight Loss | interventions — Tablets

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 (Active Comparator): High dairy intake and calcium supplement. High intake of low-fat milk product intake (3-4 servings per day) plus one 350 mg calcium supplement per day during 500 kcal/day deficit diet.
  Interventions: Behavioral: High dairy and calcium intake
- 1 (Placebo Comparator): Usual diet of low dairy and calcium intake. Usual intake of low milk product intake (1 serving/day) and low calcium intake with a placebo during a 500 kcal/day deficit diet.
  Interventions: Behavioral: Usual intake

INTERVENTIONS:
Behavioral: High dairy and calcium intake — High intake of low-fat milk product intake (3-4 servings per day) plus one 350 mg calcium supplement per day during 500 kcal/day deficit diet.
  Other Names: Jamieson Mega Cal™ Chewable Calcium (350 mg) tablet
  Arms: 2
Behavioral: Usual intake — Usual intake of low milk product intake (1 serving/day) and low calcium intake with a placebo during a 500 kcal/day deficit diet
  Arms: 1

SUMMARY:
The purpose of this study is to determine if increased intake of low-fat milk products and calcium as part of a calorie restricted diet helps achieve a healthier body weight and body composition and decrease blood glucose levels in people with insulin resistance or type 2 diabetes.

DETAILED DESCRIPTION:
Obesity can cause many health problems as it is linked to several chronic diseases including type 2 diabetes. We know that individuals who are overweight or obese, and have impaired glucose tolerance or insulin resistance, have a good chance of developing type 2 diabetes. Research tells us that the risk of developing type 2 diabetes can be decreased by losing weight and making dietary changes. A promising area of study involves using low-fat milk products and calcium to prevent and/or control obesity and diabetes. This study is important because it will determine if including low-fat milk products in weight reducing diets can enhance weight loss, improve fat loss and decrease levels of blood glucose and insulin in individuals with impaired glucose tolerance or type 2 diabetes not treated with medication. This information is directly applicable to treating diseases such as obesity, type 2 diabetes and heart disease.

ELIGIBILITY:
Inclusion Criteria:

* Overweight and obese (BMI of 27 to 37 kg/m2)
* Impaired glucose tolerance (fasting blood glucose >5.6 mmol/L) or
* Type 2 diabetes treated with diet and exercise alone (no medications)
* One or more of the following criteria for metabolic syndrome:

  1. Hypertriglyceridemia (> 1.70 mmol/L)
  2. Low high-density lipoprotein (HDL) cholesterol (< 1.04 mmol/L in men and < 1.30 mmol/L in women)
  3. High blood pressure (> 130/85 mm Hg)
  4. High waist circumference ( > 94 cm in men, > 80 cm in women)
* Weight stable and no changes in exercise in past 3 months

Exclusion Criteria:

* Type 1 diabetes
* Type 2 diabetes treated with oral hypoglycemic agents or insulin
* HbA1c > 8%
* myocardial infarction or have undergone a cardiovascular intervention within the past three months
* Subjects taking fibrate or statins who have had a dose change within the 8 weeks prior to randomization
* Liver or pancreas disease
* Major gastrointestinal surgeries
* Pregnant or lactating
* Exhibit alcohol or drug dependence
* Taking drugs influencing appetite
* Have a milk allergy or lactose intolerance
* Following a diet or exercise regime designed for weight loss
* Have a body weight greater than 350 lb (weight limit for DEXA instrument)
* Chronic use of bulk laxatives, antacids or calcium supplements

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2007-10; Primary Completion 2009-04 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Weight loss | 12 weeks

SECONDARY OUTCOMES:
Insulin and glucose response | 12 weeks
Inflammatory Markers | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Raylene A. Reimer, PhD, RD, Principal Investigator — University of Calgary
Locations (1):
- Faculty of Kinesiology, Roger Jackson Centre for Health and Wellness Research, Calgary, Alberta, Canada